CLINICAL TRIAL: NCT00151203
Title: A Phase II Study of Clarithromycin (Biaxin), Lenalidomide (Revlimid), and Dexamethasone (Decadron) for Newly Diagnosed Subjects With Multiple Myeloma
Brief Title: Phase II Study of Biaxin, Revlimid, and Dexamethasone for Untreated Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0409007427
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Multiple Myeloma
Keywords: newly diagnosed multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Clarithromycin; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Clarithromycin, Lenalidomide, Dexamethasone — Dexamethasone (Decadron®) will be given orally at a dose of 40 mg on days 1, 2, 3, 8, 15 and 22 during the first cycle and once a week on days 1, 8, 15, and 22 for each subsequent cycle.
  Clarithromycin (Biaxin®) will be given orally at a dose of 500 mg twice a day beginning on day 2 of cycle 1.
  Lenalidomide (Revlimid®) will be given orally at a dose of 25 mg daily beginning on day 3 and ending on day 21 of cycle 1 and on days 1-21 of subsequent cycles.

SUMMARY:
PRIMARY STUDY OBJECTIVES

* To evaluate the efficacy of the combination of clarithromycin (Biaxin®), lenalidomide (Revlimid™), and dexamethasone (Decadron®) as an induction therapy for patients with newly diagnosed multiple myeloma (MM).
* To evaluate the safety of the combination of clarithromycin, lenalidomide, and dexamethasone as an induction therapy for patients with newly diagnosed MM.

SECONDARY STUDY OBJECTIVES

* To examine the role of clarithromycin on the pharmacokinetic properties of dexamethasone and lenalidomide.
* To examine the angiogenesis profile in untreated patients and in patients receiving induction therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject must voluntarily sign and understand written informed consent.
* Histologically confirmed Durie-Salomon stage II or III MM (see Appendix II). Stage I MM patients will be eligible if they display poor prognostic factors (ß2M > or = 5.5 mg/L, plasma cell proliferation index > or = 5%, albumin of less then 3.0, and unfavorable cytogenetics).
* Measurable disease as defined by > 1.0 g/dL serum monoclonal protein, >0.1 g/dL serum free light chains, > 0.2 g/24 hrs urinary M-protein excretion, and/or measurable plasmacytoma(s).
* Age > or = 18 years at the time of signing the informed consent form.
* Karnofsky performance status > or = 70% (>60% if due to bony involvement of myeloma (see Appendix V).
* No prior treatment or less than one full course of first-line therapy. Patients may be receiving adjuvant antiresorptive therapy (i.e., pamidronate or zoledronic acid) as routine care.
* If the patient is a woman of childbearing age, she must have a negative serum or urine pregnancy test within 7 days of starting study.
* Due to the unknown risk of teratogenic side effects, subjects (women and men) must agree to use effective contraception throughout the duration of the study and for at least 1 month after discontinuation of study drugs.
* Life expectancy > 3 months
* Absolute neutrophil count (ANC)> or = 1000 cells/mm3 (1.0 x 109/L)
* Platelets count > or = 75,000/mm3 (75 x 109/L)
* Serum SGOT/AST < 3.0 x upper limits of normal (ULN)
* Serum SGPT/ALT < 3.0 x upper limits of normal (ULN)
* Serum creatinine < 2.5 mg/dL (221 µmol/L)
* Serum total bilirubin < 2.0 mg/dL (34 µmol/L)

Exclusion Criteria:

* Patients with non-secretory MM (no measurable monoclonal protein, free light chains, and/or M-spike in blood or urine).
* Prior history of other malignancies (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless disease free for ³ 5 years.
* NYHA Class III or IV heart disease. History of active angina, congestive heart disease, or myocardial infarction within 6 months.
* Pregnant or lactating women are ineligible.
* Known HIV positivity
* Active viral or bacterial infections or any coexisting medical problem that would significantly increase the risks of this treatment program.
* Known hypersensitivity to dexamethasone, clarithromycin, lenalidomide, or thalidomide.
* Prior therapy for the treatment of MM
* History of thromboembolic event or other condition currently requiring anticoagulation with warfarin (Coumadin). Patients whose therapy is changed to heparin are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-12 (Actual); Primary Completion 2007-04 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Response rate, time to maximum response, toxicities | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Niesvizky, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

REFERENCES:
- [Derived] Rossi A, Mark T, Jayabalan D, Christos P, Zafar F, Pekle K, Pearse R, Chen-Kiang S, Coleman M, Niesvizky R. BiRd (clarithromycin, lenalidomide, dexamethasone): an update on long-term lenalidomide therapy in previously untreated patients with multiple myeloma. Blood. 2013 Mar 14;121(11):1982-5. doi: 10.1182/blood-2012-08-448563. Epub 2013 Jan 8. PMID 23299315
- [Derived] Niesvizky R, Jayabalan DS, Christos PJ, Furst JR, Naib T, Ely S, Jalbrzikowski J, Pearse RN, Zafar F, Pekle K, Larow A, Lent R, Mark T, Cho HJ, Shore T, Tepler J, Harpel J, Schuster MW, Mathew S, Leonard JP, Mazumdar M, Chen-Kiang S, Coleman M. BiRD (Biaxin [clarithromycin]/Revlimid [lenalidomide]/dexamethasone) combination therapy results in high complete- and overall-response rates in treatment-naive symptomatic multiple myeloma. Blood. 2008 Feb 1;111(3):1101-9. doi: 10.1182/blood-2007-05-090258. Epub 2007 Nov 7. PMID 17989313